CLINICAL TRIAL: NCT01289977
Title: Immune Responses After Human Subject Challenge With Sand Fly Bites: Exploratory Study for Selection of Potential Leishmania Vaccine Antigen Candidates
Brief Title: Immune Responses After Human Subject Challenge With Sand Fly Bites
Status: Completed | Type: Observational
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: G183ZU; Y1-AI-0744-01 (Other Grant/Funding Number: NIAID Interagency Agreement)
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: Sandfly; leishmaniasis; immune response; individuals age 18-50
MeSH Terms: conditions — Leishmaniasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and white blood cells will be retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Phlebotomus group: Those in the Phlebotomus group will have exposure to P. duboscqui sand fly
- Lutzomyia group: Those placed in this group will receive exposure to L. longipalpis sand fly bites.

SUMMARY:
Sand flies can carry the infection leishmaniasis (a parasite). The purpose of this study is to evaluate the human immune response to uninfected laboratory raised sand fly bites and select from the immune response to sand fly saliva, possible substances to use for a future vaccine to protect against the parasite leishmaniasis.

DETAILED DESCRIPTION:
Based on travel history and possible exposure, subjects were entered into one of 2 arms, Ph. dubosqui or Lu. lutzomyia controlled sand fly repeated feedings. At baseline a pheresis was done to collect baseline cells. Subjects received sand fly bites on a q2 week schedule for 2 months followed by a q2 months schedule for one year. They had an option to extend for a late recall feeding at 18 months, when a skin biopsy was performed 48 hours after sand fly bites. Currently the study is fully enrolled and all human subject contact is complete. We (laboratory at NIAID) are studying the humoral, cellular immune responses using blood samples, and cytokine expression in the skin biopsy samples.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Plans to remain in DC area for at least one year
* willingness to participate in all study procedures
* general good health
* military health care beneficiary
* able to provide informed consent

Exclusion Criteria:

* Prior travel to geographic areas where leishmania transmitting sand flies are common
* positive antibody to sand fly saliva on screening blood test
* pregnancy
* elevated serum IgE
* history of chronic medical illness
* adult history of treatment requiring anemia
* large reactions to insect bites
* history of multiple vasovagal reactions to phlebotomy
* difficult venous access for phlebotomy
* Taking medications that could interfere with immune responses

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male and female military health care beneficiaries in good health, age 18-50
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2010-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04-15 (Actual)

PRIMARY OUTCOMES:
Human Th1 immune response to specific sand fly salivary proteins | 6-18 months
  Subject blood will be obtained at set points after repeated controlled sand fly feedings, duration for 20 minutes. Sand fly salivary molecules that demonstrate a strong Th1 immune response in these human PBMC, and little Th2 cytokine induction will be considered for development as future leishmania vaccine antigen candidates.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi E Aronson, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States